CLINICAL TRIAL: NCT04905290
Title: Conduction System Pacing Optimized Therapy Study
Brief Title: Conduction System Pacing Optimized Therapy
Acronym: CSPOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT20029
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Results first posted 2025-01-17 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2023-10

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single Arm (Experimental): Patients will undergo 1) Conduction System Pacing Optimized Therapy (CSPOT) lead placement, then the 2) acute pacing protocol, and then 3) device implant. During the acute pacing protocol (step 2), all patients will undergo three types of pacing configurations and for each pacing configuration several delay settings, as defined in Assigned Interventions. For each intervention, defined as a unique combination of pacing configuration and delay setting, the protocol will alternate for several heartbeats between AV pacing and intervention (5 sections of AV pacing and 4 sections of intervention). For each set of 9, Left Ventricular dP/dt max will be calculated continuously, and Standard Deviation of Activation Time will be selected from one of the sections for atrial-only pacing and one of the intervention sections. Device implant (step 3) will be with either a CRT-D or CRT-P. Each patient's device will be programmed to CSPOT pacing. Patients will be followed for 6 months.
  Interventions: Device: Left ventricular coronary sinus (BiV) configuration; Device: Conduction system pacing-only configuration; Device: Conduction System Pacing Optimized Therapy (CSPOT) configuration

INTERVENTIONS:
Device: Left ventricular coronary sinus (BiV) configuration — For subjects with a pacemaker, pacing of the left ventricular coronary sinus only. For subjects with a defibrillator, biventricular pacing of the left ventricular coronary sinus and the right ventricle. During the acute protocol, the five AV delays for this intervention include the default AV delay setting, default + 30 milliseconds (ms) AV delay, default + 60 ms AV delay, default - 30ms AV delay, default - 60ms AV delay. Patients with a defibrillator will receive two additional delays LV precedes default by 30ms and LV precedes default by 60ms.
Device: Conduction system pacing-only configuration — Conduction System Pacing (CSP) of the left bundle branch. During the acute protocol, the five AV delays for this intervention include the default AV delay setting, default + 30 milliseconds (ms) AV delay, default + 60 ms AV delay, default - 30ms AV delay, and default - 60ms AV delay.
Device: Conduction System Pacing Optimized Therapy (CSPOT) configuration — A combination of Left Ventricle pacing and Conduction System Pacing of the left bundle branch. During the acute protocol, the eight delays for this intervention include the default AV delay setting, default + 30 milliseconds (ms) AV delay, default + 60 ms AV delay, default - 30ms AV delay, default - 60ms AV delay, CSP precedes default by 30ms, LV precedes default by 30ms and LV precedes default by 60ms.

SUMMARY:
The purpose of the CSPOT study is to determine the best mode of cardiac resynchronization therapy (CRT) pacing for different populations of CRT patients, comparing traditional biventricular or left ventricular pacing (BiV), conduction system pacing (CSP)-only, and conduction system pacing optimized therapy (CSPOT) also known as a combination of conduction system pacing (CSP) and left ventricular (LV) pacing. Additionally, safety of the system will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to provide written informed consent
* Subject is at least 18 years of age
* Patient is willing and able to comply with the protocol, including follow-up visits
* The patient's medical records must be accessible by the enrolling site over the follow-up period
* Standard CRT-D or CRT-P indications, with a preference for IVCD and non-LBBB patients, where LBBB is defined according to Strauss criteria.
* De-novo CRT implant, including upgrade from pacemaker or ICD

Exclusion Criteria:

* Subject has persistent or permanent AF (Atrial Fibrillation)/AFL (Atrial Flutter)
* Subject has 2nd or 3rd degree AV (Atrioventricular) Block
* Subject has RBBB with no additional conduction block
* Subject has intrinsic (non-paced) QRS width less than or equal to 120 ms
* Subject experienced MI within 40 days prior to enrollment
* Subject underwent valve surgery, within 90 days prior to enrollment
* Subject is post heart transplantation or is actively listed on the transplantation list
* Subject is implanted with a LV assist device
* Subject has severe renal disease
* Subject is on continuous or uninterrupted infusion (inotropic) therapy for heart failure
* Subject has severe aortic stenosis (with a valve area of <1.0 cm or significant valve disease expected to be operated within study period)
* Subject has severe aortic calcification or severe peripheral arterial disease
* Subject has complex and uncorrected congenital heart disease
* Subject has mechanical heart valve
* Pregnant or breastfeeding woman (pregnancy test required for woman of child-bearing potential and who are not on a reliable form of birth regulation method or abstinence)
* Subject is enrolled in another study that could confound the results of this study without documented pre-approval from Medtronic study manager

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-27 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-11-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (7):
  - University of South Florida, Tampa, Florida
  - The University of Chicago Medicine, Chicago, Illinois
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Medtronic Inc, Mounds View, Minnesota
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Beacon Hospital, Dublin, Ireland
- Poland (2):
  - Górnośląskie Centrum Medyczne im prof Leszka Gieca Śląskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - Szpital Uniwersytecki w Krakowie, Krakow
- United Kingdom (2):
  - Hammersmith Hospital, London
  - Great Western Hospital, Swindon

REFERENCES:
- [Derived] Jastrzebski M, Foley P, Chandrasekaran B, Whinnett Z, Vijayaraman P, Upadhyay GA, Schaller RD, Gardas R, Richardson T, Kudlik D, Stadler RW, Zimmerman P, Burrell J, Waxman R, Cornelussen RN, Lyne J, Herweg B. Multicenter Hemodynamic Assessment of the LOT-CRT Strategy: When Does Combining Left Bundle Branch Pacing and Coronary Venous Pacing Enhance Resynchronization?: Primary Results of the CSPOT Study. Circ Arrhythm Electrophysiol. 2024 Nov;17(11):e013059. doi: 10.1161/CIRCEP.124.013059. Epub 2024 Oct 23. PMID 39440428

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 60
Implant Attempt | 55
Completed | 42
Not Completed | 18
Not completed — Adverse Event | 4
Not completed — Death | 2
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 2
Not completed — Screen Failure | 2
Not completed — Unsuccessful Procedure | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 39
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 18
  More than one race | 0
  Unknown or Not Reported | 38
Height [Mean (Standard Deviation); unit: cm] | 171.1 (10.5)
Weight [Mean (Standard Deviation); unit: kg] | 88.2 (18.9)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 121.9 (17.5)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 70.8 (10.4)
NYHA Classification [Count of Participants; unit: Participants] — Class I:No symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  Class II:Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  Class III:Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m).Comfortable only at rest.
  Class IV:Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  No NYHA class listed or unable to determine. Lower scores have less severe heart failure.
  Participants
    Class I | 5
    Class II | 29
    Class III | 24
    Class IV | 1
    Not Available | 1

OUTCOME MEASURES:

1. Primary Outcome: Electrical Synchronization Response
Description: Standard Deviation of Activation Times (SDAT) is a measurement of dyssynchrony, taken by the ECG belt. As described in the SDAT Acute Protocol (below) and intervention sections, percent change in SDAT from AV-only pacing was calculated for each patient-pacing configuration combination over the 5 AV delays. Within each patient the difference between CSPOT SDAT and CSP SDAT and the difference between CSPOT SDAT and BiV SDAT were taken. The mean of those differences across patients was calculated along with a 95% confidence interval.
Time Frame: At implant during acute protocol
Population: Subjects with SDAT measurements available for each pacing configuration.
Measure: Mean (95% Confidence Interval); unit: Difference in percent change in SDAT
Groups:
- SDAT Acute Protocol: For each intervention, data from 9 sections of atrial only pacing and intervention will be used, beginning with the atrial-only pacing that immediately precedes the first intervention section and ending with the atrial-only pacing immediately following the last intervention pacing section. The SDAT measurement will be taken during one of the 4 intervention pacing sections and one of the 5 atrial-only pacing sections. This will provide 1 pair of SDAT measurements for each patient-intervention combination. For each pair, the percent change from the atrial-only section to the intervention section will be computed. Within each patient, the percent changes calculated from the 5 AV delay settings (default, default + 30ms, default + 60ms, default - 30ms, default - 60ms) will be used to fit a quadratic curve. The minimum value from the fitted quadratic curve within the delay settings will be used as the SDAT measurement for that patient-pacing configuration combination.
Arm/Group | SDAT Acute Protocol
Number analyzed (Participants) | 44
Difference in percent change in SDAT
  CSPOT vs CSP | 15.18 [4.26 to 26.09]
  CSPOT vs BiV | 17.04 [4.32 to 29.76]

2. Primary Outcome: Hemodynamic Response
Description: Left Ventricular (LV) dP/dt max, a measurement of the initial velocity of myocardial contraction. As described in the LV dP/dt max (below) and intervention sections, percent change in LV dP/dt max from AV-only pacing was calculated for each patient-pacing configuration combination over the 5 AV delays. Within each patient the difference between CSPOT SDAT and CSP SDAT and the difference between CSPOT SDAT and BiV SDAT were taken. The mean of those differences across patients was calculated along with a 95% confidence interval.
Time Frame: At implant during acute protocol
Population: Subjects with LV dP/dt max measurements available for each pacing configuration
Measure: Mean (95% Confidence Interval); unit: Difference in % change LV dP/dt max
Groups:
- LV dP/dt Max Acute Protocol: For each intervention, data from 9 sections of atrial only pacing and intervention will be used, beginning with the atrial-only pacing that immediately precedes the first intervention section and ending with the atrial-only pacing immediately following the last intervention pacing section. For each of the nine sections, the section will be split into the "first half" and "second half". For each half section, the median of the LV dP/dt max values for beats within the defined period will be calculated. This will provide eight pairs of medians from adjacent atrial-only pacing and intervention-delay setting combination sections. For each pair, the percent change from the atrial-only section median to the intervention section median will be computed. This will be repeated for each delay setting described in the intervention section. Within each patient, the median percent changes calculated from the 5 AV delay settings (default, default + 30ms, default + 60ms, default - 30ms, default - 60ms) will be used to fit a quadratic curve. The maximum value from the fitted quadratic curve within the delay settings will be used as the LV dP/dt max measurement for that patient-pacing configuration combination.
Arm/Group | LV dP/dt Max Acute Protocol
Number analyzed (Participants) | 41
Difference in % change LV dP/dt max
  CSPOT vs CSP | 10.33 [7.15 to 13.51]
  CSPOT vs BiV | -1.31 [-4.75 to 2.13]

3. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Left ventricular ejection fraction will be measured, based on echocardiography, at the baseline visit and again at the 6-month follow-up visit. Change will be calculated as the value observed at baseline subtracted from the value observed at 6 months.
Time Frame: Baseline and 6 months
Population: Subjects with LVEF measurements at both baseline and 6-month follow-up visit
Measure: Mean (95% Confidence Interval); unit: Change in percentage of LVEF
Arm/Group | Single Arm
Number analyzed (Participants) | 35
Change in percentage of LVEF | 15.24 [10.16 to 20.32]

4. Secondary Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: Left ventricular end systolic volume will be measured, based on echocardiography, at the baseline visit and again at the 6-month follow-up visit. The change will be calculated as difference between the 6-month and baseline values, divided by the baseline value.
Time Frame: Baseline and 6 months
Population: Subjects who had LVESV recorded at both baseline and the 6-month follow-up visit
Measure: Mean (95% Confidence Interval); unit: percent change lvesv
Arm/Group | Single Arm
Number analyzed (Participants) | 35
percent change lvesv | -43.28 [-51.51 to -35.06]

5. Secondary Outcome: Clinical Composite Score (CCS)
Description: The Clinical Composite Score (CCS) is a validated 3-level categorical variable that can take the values - Improved, Unchanged, or Worsened - at each follow-up visit. It is based on mortality, HF events, termination of device function, NYHA score, and patient global assessment. Briefly, the scoring system is as follows:
  * A patient is considered "worsened" if they die, demonstrate a worsened NYHA class, report at least moderately worsened heart-failure symptoms, or are hospitalized or permanently discontinue therapy because of or associated with worsening heart-failure
  * A patient is considered "improved" if they have not "worsened" and either demonstrate improvement in NYHA class or report at least moderately improved heart-failure symptoms
  * A patient is considered "stabilized" if they have not "worsened" or "improved"
  * A patient is considered "unavailable" if they did not complete 6-month visit and was not "worsened"
Time Frame: 6 months
Population: Subjects who had a successful implant procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 46
Participants
  Improved | 35
  Stabilized | 2
  Worsened | 6
  Unavailable | 3

6. Secondary Outcome: Absolute Percent Change in SDAT by QRS Subgroup
Description: Percent change in SDAT (as described in Primary Outcome 1: Arm/Group Description) by baseline QRS subgroup for each pacing configuration CSP, BiV, CSPOT during acute protocol at implant.
  The QRS subgroups were subjects with QRS width greater than 171ms and QRS width less than or equal to 171ms as measured by 12-lead ECG
Time Frame: At Implant during acute protocol
Population: Subjects who had SDAT measured during the acute protocol.
Measure: Mean (95% Confidence Interval); unit: abs percent change in SDAT
Groups:
- QRS Greater Than 171ms: Subjects who completed acute protocol with QRS width greater than 171ms as measured by 12-lead ECG. SDAT
- QRS Less Than or Equal to 171ms: Subjects who completed acute protocol with QRS width less than or equal to 171ms as measured by 12-lead ECG
Arm/Group | QRS Greater Than 171ms | QRS Less Than or Equal to 171ms
Number analyzed (Participants) | 24 | 24
abs percent change in SDAT
  CSPOT: number analyzed (Participants) | 20 | 24
  CSPOT | 42.77 [30.21 to 55.32] | 42.46 [31.6 to 53.32]
  BIV: number analyzed (Participants) | 22 | 24
  BIV | 34.61 [23.94 to 45.28] | 19.72 [-7.96 to 47.41]
  CSP | 34.26 [26.1 to 42.42] | 22.05 [-2.18 to 46.28]

7. Secondary Outcome: Absolute Percent Change in SDAT Split by Subjects With Pure LBBB and With Other Conduction Disorders
Description: Percent change in SDAT (as described in Primary Outcome 1: Arm/Group Description) split by subjects with pure Left Bundle Branch Block (LBBB) and with other Conduction Disorders for each pacing configuration CSP, BiV and CSPOT during acute protocol.
Time Frame: At Implant during acute protocol
Population: Subjects who had SDAT measured during the acute protocol.
Measure: Mean (95% Confidence Interval); unit: abs percent change in SDAT
Groups:
- LBBB: Subjects who completed acute protocol and had pure Left Bundle Branch Block
- NIVCD: Subjects who completed acute protocol who had conduction disorder other than pure Left Bundle Branch Block
Arm/Group | LBBB | NIVCD
Number analyzed (Participants) | 19 | 29
abs percent change in SDAT
  CSPOT: number analyzed (Participants) | 15 | 29
  CSPOT | 51.47 [41.44 to 61.5] | 38.01 [27.22 to 48.79]
  BIV: number analyzed (Participants) | 17 | 29
  BIV | 36.28 [28.36 to 44.2] | 21.31 [-2.24 to 44.87]
  CSP | 40.18 [33.91 to 46.44] | 20.28 [0.14 to 40.42]

8. Secondary Outcome: Absolute Percent Change in SDAT Split by Subjects With Ischemic Cardiomyopathy and Those With Non-Ischemic Cardiomyopathy
Description: Absolute Percent change in SDAT (as described in Primary Outcome 1: Arm/Group Description) split by subjects with Ischemic Cardiomyopathy and those with Non-Ischemic Cardiomyopathy for each pacing configuration CSP, BiV and CSPOT during acute protocol.
Time Frame: At Implant during acute protocol
Population: Subjects who had SDAT measured during the acute protocol.
Measure: Mean (95% Confidence Interval); unit: abs percent change in SDAT
Groups:
- Non-Ischemic: Subjects who completed acute protocol and had Non-Ischemic Cardiomyopathy
- Ischemic: Subjects who completed acute protocol who had Ischemic Cardiomyopathy
Arm/Group | Non-Ischemic | Ischemic
Number analyzed (Participants) | 34 | 14
abs percent change in SDAT
  CSPOT: number analyzed (Participants) | 30 | 14
  CSPOT | 48.96 [41.32 to 56.61] | 28.95 [10.75 to 47.15]
  BIV: number analyzed (Participants) | 32 | 14
  BIV | 36.95 [29.71 to 44.20] | 3.74 [-44.37 to 51.85]
  CSP | 38.83 [32.17 to 45.49] | 2.23 [-37.24 to 41.71]

9. Secondary Outcome: Percent Change in LV dP/dt Max Split by Subjects With Ischemic Cardiomyopathy and Those With Non-Ischemic Cardiomyopathy
Description: Percent change in LV dP/dt max (as described in Primary Outcome 2: Arm/Group Description)split by subjects with Ischemic Cardiomyopathy and those with Non-Ischemic Cardiomyopathy for each pacing configuration CSP, BiV and CSPOT during acute protocol.
Time Frame: At Implant during acute protocol
Population: Subjects who had LV dP/dt max measured during acute protocol
Measure: Mean (95% Confidence Interval); unit: percent change in LV dP/dt max
Arm/Group | Non-Ischemic | Ischemic
Number analyzed (Participants) | 31 | 14
percent change in LV dP/dt max
  CSPOT: number analyzed (Participants) | 27 | 14
  CSPOT | 30.05 [23.81 to 36.29] | 17.56 [10.82 to 24.31]
  BIV: number analyzed (Participants) | 29 | 14
  BIV | 30.64 [22.15 to 39.12] | 17.62 [11.56 to 23.69]
  CSP | 20.03 [15.96 to 24.1] | 8.32 [2.13 to 14.51]

10. Secondary Outcome: Percent Change in LV dP/dt Max Split by Subjects With Pure Left Bundle Branch Block (LBBB) and With Other Conduction Disorders (NIVCD)
Description: Percent change in LV dP/dt max (as described in Primary Outcome 2: Arm/Group Description) split by subjects with pure Left Bundle Branch Block (LBBB) and with other Conduction Disorders (NIVCD) for each pacing configuration CSP, BiV and CSPOT during acute protocol
Time Frame: At Implant during acute protocol
Population: Subjects who had LV dP/dt max measured during acute protocol
Measure: Mean (95% Confidence Interval); unit: percent change in LV dP/dt max
Arm/Group | LBBB | NIVCD
Number analyzed (Participants) | 18 | 27
percent change in LV dP/dt max
  CSPOT: number analyzed (Participants) | 14 | 27
  CSPOT | 28.08 [20.4 to 35.76] | 24.59 [17.98 to 31.21]
  BIV: number analyzed (Participants) | 16 | 27
  BIV | 29.35 [17.73 to 40.98] | 24.65 [17.05 to 32.25]
  CSP | 18.02 [12.65 to 23.39] | 15.29 [10.12 to 20.47]

11. Secondary Outcome: Improvement in LV dP/dt Max by QRS Subgroup
Description: Percent change in LV dP/dt max (as described in Primary Outcome 2: Arm/Group Description) by QRS subgroup for each pacing configuration CSP, BiV and CSPOT during acute protocol. The QRS subgroups were subjects with QRS width greater than 171ms and QRS width less than or equal to 171ms as measured by 12-lead ECG
Time Frame: At Implant during acute protocol
Population: Subjects who had LV dP/dt max measured during acute protocol
Measure: Mean (95% Confidence Interval); unit: percent change in LV dP/dt max
Groups:
- QRS Greater Than 171ms: Subjects who completed acute protocol with QRS width greater than 171ms as measured by 12-lead ECG
Arm/Group | QRS Greater Than 171ms | QRS Less Than or Equal to 171ms
Number analyzed (Participants) | 23 | 22
percent change in LV dP/dt max
  CSPOT: number analyzed (Participants) | 19 | 22
  CSPOT | 29.28 [21.32 to 37.24] | 22.77 [16.39 to 29.14]
  BIV: number analyzed (Participants) | 21 | 22
  BIV | 32.18 [20.68 to 43.68] | 20.88 [15.74 to 26.02]
  CSP | 18.2 [12.88 to 23.51] | 14.49 [9.16 to 19.82]

ADVERSE EVENTS:
Time Frame: From enrollment through 6 month follow-up
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 2/60
Serious Adverse Events (participants affected / at risk) | 20/60
Other Adverse Events (participants affected / at risk) | 14/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=60)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Cardiac perforation (Cardiac disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Device fastener issue (Product Issues) | 1 (1)
Device lead issue (Product Issues) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=60)
Atrial fibrillation (Cardiac disorders) | 5 (5)
Atrioventricular block complete (Cardiac disorders) | 3 (4)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (2)
Adrenal mass (Endocrine disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Implant site haematoma (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 2 (2)
Peripheral swelling (General disorders) | 1 (1)
Device placement issue (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site swelling (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Device stimulation issue (Product Issues) | 2 (2)
Lead dislodgement (Product Issues) | 1 (1)
Oversensing (Product Issues) | 2 (2)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/90/NCT04905290/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-02): https://cdn.clinicaltrials.gov/large-docs/90/NCT04905290/SAP_002.pdf